CLINICAL TRIAL: NCT05603533
Title: The Effectiveness of a Music and Video-based Group Exercise Therapy in Older Adults With Moderate Dementia
Brief Title: Adherence by Music to Exercise in Dementia: Group Therapy
Acronym: AMUSED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Stichting Alzheimer Onderzoek (Unknown)
Responsible Party: Principal Investigator, Tinne Plattiau, Msc, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMUSED STUDY 1
Record Dates: First submitted 2022-10-20; First posted 2022-11-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Dementia
Keywords: Exercise therapy; Rehabilitation; Physical therapy; Frailty; Treatment Adherence and Compliance; Cognition; Physical functioning
MeSH Terms: conditions — Dementia; Frailty; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): On top of the regular physical therapy, the participants in the intervention group will receive a music and video-based group exercise therapy in small groups of 5. On a big screen, a video of an older woman performing exercises will be shown, the participants will have to copy these exercises. In the beginning of each session, the participants will be able to choose the music they want to move to.
  Interventions: Other: Music and video-based group exercise therapy
- Control group (No Intervention): The participants in the control group will receive no additional therapy.

INTERVENTIONS:
Other: Music and video-based group exercise therapy — Each exercise session will last up to 45min. The participants will follow this group exercise therapy twice a week for four months.
  Arms: Intervention group

SUMMARY:
The aim of this study is to asses the effect of a music and video-based group exercise therapy on motivation, physical functioning, cognition and well-being in older adults with moderate dementia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with moderate dementia (MMSE between 12 and 20)
* Age 65 years or older
* Resident in nursing home for at least 30 days
* Able to stand (supported) for 10 seconds with supervision

Exclusion Criteria:

* Inadequate functional hearing
* Uncorrected visual problems
* Rehabilitating from an orthopedic or neurologic insult
* Known disability that significantly influences 6 month prognosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The change in motivation between 1,2,3 and 4 months into the intervention will be measured using the observed emotion rating scale (OERS) | 1,2,3 and 4 months of intervention
  The OERS evaluates the positive (pleasure, interest/alertness) and negative mood (anger, anxiety, sadness) by observing the extent or duration of facial expressions and body movements and has a moderate to high interrater reliability. To evaluate the OERS, two exercise sessions will be recorded each month and results will be averaged to compensate for daily fluctuations.
The change in muscle strength between baseline, mid-intervention and at the end of intervention will be measured using the modified timed chair stand test. | At baseline, after 2 and 4 months
  The timed chair stand test is a valid and reliable test to evaluate muscle strength in older adults. The participant will be asked to stand up and sit back down on a chair five times without using their hands. The time it takes to perform this task will be measured.
The change in muscle strength between baseline, mid-intervention and at the end of intervention will be measured using a hand-held dynamometer | At baseline, after 2 and 4 months
  When using the hand-held dynamometer to measure strength, the break technique will be used. The examiner will apply resistance in a fixed position and the person being tested exerts a maximum effort against the dynamometer for 3-5 seconds. At the last second, the examiner applies a resistance sufficient to overcome the maximum effort of the person being tested and cause the subject's joint to move.
The change in compliance between 1,2,3 and 4 months into the intervention will be measured | 1,2,3 and 4 months of intervention
  Compliance will be measured by assessing whether the participants exercised at the prescribed intensity. To evaluate compliance, two exercises sessions will be recorded and results will be averaged to compensate for daily fluctuations. Both quality and quantity of the participants' performances will be scored. To measure the quantity, the amount of repetitions the participant performed will be rated from zero (no repetitions) to three (all repetitions). A score of two was chosen as cut-off score, indicating that more than half of the exercises were performed. To measure quality, the recorded performances will be compared with the visual instructions on the TV-screen and will be scored on a scale from zero (no repetitions) to three (the performance matched completely with the instructions). A score of two was chosen as cut-off score, indicating that more than half of the exercises were matched with the instructions.
The change in adherence between 1,2,3 and 4 months into the intervention will be measured | 1,2,3 and 4 months of intervention
  Adherence will be measured by counting the amount of therapy sessions each participant completed (%)
Attrition rate | Twice a week for 4 months
  The amount of participants that discontinued the program

SECONDARY OUTCOMES:
The change in balance and gait between baseline, mid-intervention and at the end of intervention will be measured using the Tinetti test | At baseline, after 2 and 4 months
  The Tinetti test was developed to assess gait and balance in older adults and to assess perception of balance and stability during activities of daily living and fear of falling. It's also used as an indicator of the fall risk of an individual. During the test, the participant will be asked to perform certain tasks. The examiner will look at certain key points to score these tasks.
The change in activity level and sleep between baseline, mid-intervention and at the end of intervention will be measured using an Actigraph | At baseline, after 2 and 4 months
  The actigraph is a validated, 3 axis accelerometer that will be used to measure activity level (inactivity/sedentary behavior as well as general restlessness and wandering behavior) and sleep. The device will be worn for five consecutive days. During the day, the actigraph will be worn at the hip to measure activity and during the night, the actigraph will be worn at the wrist to measure sleep.
The change in cognition between baseline, mid-intervention and at the end of intervention will be assessed using the Montreal Cognitive Assessment (MOCA) | At baseline, after 2 and 4 months
  The MoCA is a tool used to determine if cognitive impairment is present. It takes around ten minutes to complete. It evaluates visuospatial skills, attention, language, abstract reasoning, delayed recall, executive function, and orientation.
The change in quality of life between baseline, mid-intervention and at the end of intervention will be assessed using the ICEpop CAPability measure for Older people (ICECAP-O) | At baseline, after 2 and 4 months
  The ICECAP-O questionnaire is validated self-report measure for quality of life in older adults with mild and moderate dementia. The ICECAP-O focuses on a broader sense of wellbeing, rather than only health related quality of life. The measure covers attributes of wellbeing that were found to be important to older adults.
The change in behavioral and psychological symptoms of dementia between baseline, mid-intervention and at the end of intervention will be evaluated using the Dutch version of the Cohen-Mansfield Agitation Inventory (CMAI-D) | At baseline, after 2 and 4 months
  The CMAI-D is a 29-item scale to assess agitation. The participants are rated by the staff of the nursing home regarding the frequency with which, over the past two weeks, they manifested agitated behaviors. Each item is rated on a 7-point scale ranging from "Never" to "Several times per hour".

CONTACTS AND LOCATIONS:
Overall Officials: Joke Spildooren, Prof. dr., Study Director — Hasselt University
Locations (4):
- Belgium (4):
  - Aquamarijn, Kasterlee, Antwerpen
  - Woonzorgcentrum Beversthuis, Beverst, Limburg
  - Woonzorgcentrum St.Elisabeth, Hasselt, Limburg
  - Woonzorgcentrum Kimpenhof, Opglabbeek, Limburg

IPD SHARING:
Plan to Share IPD: Yes
Relevant data will be shared among collaborating researchers within Hasselt University via Google Drive. Within Google Drive, there is a division into 3 categories for access rights to personal data. To category 1 belongs only the responsible local researcher who has access to all personal data, including the log of subjects with the link between the identity and the encrypted data. To category 2 belong all employees of the research team. They have access to the pseudonymized data. To category 3 belong the master's thesis students. They only have access to the pseudonymized data relevant to their master's thesis.